CLINICAL TRIAL: NCT03722056
Title: Gastrointestinal Stromal Tumor of Stomach: Feasibility of Laparoscopic Resection in Large Lesions and Its Long Term Outcomes- A Case Series
Brief Title: Laparoscopic Management of Gastrointestinal Stromal Tumor of Stomach
Status: Completed | Type: Observational
Sponsor: GEM Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Bhushan Chittawadagi, principal investigator, GEM Hospital & Research Center
Other Study IDs: Gem/2018/1157
Record Dates: First submitted 2018-10-21; First posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Gastric GIST; Submucosal Tumor of Stomach
Keywords: Gastric GISTs; Submucosal tumours; Benign gastric lesions; Laparoscopic wedge resection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- gastric GIST: patients with suspected gastric GIST with size > 2cm are subjected for laparoscopic resection.
  Interventions: Procedure: Laparoscopic resection

INTERVENTIONS:
Procedure: Laparoscopic resection — all patients with suspected Gastric GIST undergoes laparoscopic resection. Tumour location decides the approach used for resection. Therefore, a variety of options such as local resections, wedge resections, transgastric resections, intragastric resection and partial gastrectomies were performed.

SUMMARY:
Gastric GISTs are rare neoplasms that require excision for cure. Although the feasibility of laparoscopic resection of gastric GIST less than 2cms has been established, the feasibility, safety and long-term efficacy of these techniques for larger lesions are unclear. Investigators hypothesized that laparoscopic resection of gastric GISTs even for larger lesions is feasible & results in low perioperative morbidity and an effective long-term control of the disease.

DETAILED DESCRIPTION:
Open surgical resection was the standard of treatment until two decades ago, but with advent laparoscopy and experienced gained over the years, the safety & feasibility of laparoscopic resections of gastric GISTs has been proven but for tumors less than 2 cm. However, with gain of experience and skill in laparoscopic surgery, many surgeons have reported a safety & feasibility excision of tumors greater than 5 cm. Our current study demonstrates the oncologic safety of the laparoscopic approach even with tumour size range up to 12cm, with efficacy and recurrence rates similar or superior to historical open surgical controls, however, it requires considerable expertise for safe manipulation of the tumour. All these resections were accomplished with minimal morbidity, no perioperative mortality, and short post-operative stay and comparable long term oncological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Gastric GIST>2cm size

Exclusion Criteria:

* Metastatic GIST, not fit for GA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients with suspected Gastric GIST with size more than 2 cm
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
rates of intraoperative tumour rupture | intraoperative
  Any instances of tumour rupture during surgery is noted.

CONTACTS AND LOCATIONS:
Overall Officials: sandeep sabnis, DNB SGE, Study Director — Gem Hospital & research Centre

IPD SHARING:
Plan to Share IPD: No
Data is confidential

REFERENCES:
- [Result] Keung EZ, Raut CP. Management of Gastrointestinal Stromal Tumors. Surg Clin North Am. 2017 Apr;97(2):437-452. doi: 10.1016/j.suc.2016.12.001. PMID 28325196
- [Result] Park JJ. Long-Term Outcomes after Endoscopic Treatment of Gastric Gastrointestinal Stromal Tumor. Clin Endosc. 2016 May;49(3):232-4. doi: 10.5946/ce.2016.052. Epub 2016 May 19. PMID 27196737